CLINICAL TRIAL: NCT03784469
Title: Effectiveness of Positioning on Back Pain After Transcatheter Arterial Chemoembolization Among Patients With Hepatocellular Carcinoma
Brief Title: Effectiveness of Positioning on Back Pain After TACE Among Patients With HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201712022RIND
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2018-02

CONDITIONS: Liver Cancer; Transcatheter Arterial Chemoembolization
Keywords: Transcatheter Arterial Chemoembolization; position change; back pain
MeSH Terms: conditions — Liver Neoplasms; Back Pain | interventions — Beds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Changing body position in bed (Experimental): The first hour:Supine position. The second hour:lateral position (right or left). The third hour:Supine position. The fourth hour:lateral position (right or left).
  Interventions: Other: Changing body position in bed
- Control group (No Intervention): No changing body position in bed,remaining supine position in complete bed rest and immobilized for four hours.

INTERVENTIONS:
Other: Changing body position in bed — The first hour:Supine position. The second hour:lateral position (right or left). The third hour:Supine position. The fourth hour:lateral position (right or left).
  Arms: Changing body position in bed

SUMMARY:
Changing patients' position in the bed after TACE can decrease the level of back pain without increasing the amount of bleeding and hematoma,bring patients some comfort and relieving abdominal bloating, increase patients' satisfaction.

DETAILED DESCRIPTION:
Background：During the treatment for the liver cancer patients who are treated by Transcatheter Arterial Chemoembolization (TACE), the embolic agent with chemotherapeutic drugs are injected through a catheter into a femoral artery directly supplying the tumor. Hence, after the procedure, to avoid bleeding and hematoma at the puncture site, the puncture site at groin needs to be pressed by sandbag and the affected limb needs to remain straight. These patients have to lay down on beds and are not allowed to move for at least 4 hours. Due to pressure exerted continuously to the same muscles, may cause back muscle rigidity and spasms, these patients may suffer from back pain and discomfort. In addition to usual pharmacological treatment, nursing intervention aimed at decreasing patient discomfort, therefore, this study will refer to the previous researches to develop the methods and procedures of changing body positions and apply these methods to the liver cancer patients who are treated by TACE.

Purpose：The aim of this study was to compare the level of back pain and on the amount of bleeding and hematoma between those patients changing body positions in bed and those patients not changing body positions after TACE.

Methods: This study was a randomized clinical trial. The sample consisted of 78 patients who had undergone TACE via the femoral artery, patients by using a convenience sampling assigned to either the control or experimental group (each group consisting 39 participants). All patients need to be pressed on the puncture site at groin with a sand bag of 2.5 kg for 2 hours and lie down for 4 hours. The control group received the usual care, remaining supine position in complete bed rest and immobilized. Experimental group patients received position changes in the second hour and the fourth hour after TACE.

Results: The overall trend of back pain is different between the two groups ( p <.001) , the mean of pain intensity in the second ( p =.006) and the forth hour ( p <.001) showed a significant difference. Experimental group patients had significantly less back pain than the control group after TACE . For the within subjects factor of time, the levels of back pain differed significantly across the five-time periods in experimental group ( p < .05) . In the aspect of post embolization syndrome , control group patients had significantly abdominal bloating than the experimental group ( p =.003) . None of patients developed hematoma, there was no significant difference between the two groups in terms of amount of bleeding. On the whole, experimental group patients had significantly higher satisfaction than the control group ( p =.018).

ELIGIBILITY:
Inclusion Criteria:

1. Patient with hepatocellular carcinoma hospitalized for TACE .
2. Age ≧ 18.
3. Consciousness can be communicated in Mandarin and Taiwanese.

Exclusion Criteria:

1. Symptoms of back pain before TACE.
2. Under the treatment of analagesics within 24 hours before TACE.
3. Anticoagulant was not discontinued for at least 7 days before TACE.
4. Inguinal hemorrhage or hematoma during the TACE or before removal of the vascular sheath.
5. Hemological diseases that are prone to bleeding, i.e. hemophilia and leukemia.
6. Platelet count lower than 70K or INR (international normalized ratio) is greater than 1.4.
7. No hemostatic cotton use.
8. Can not change the position in bed after TACE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
The overall trend of back pain | Within 4 hours after TACE
  The patients were asked to describe their back pain and rate its severity by using the Numerical Rating Scale (NRS-11).To determine if there is any significant difference the two groups. The NRS-11 with scores of 0 and 10 indicating no pain and excruciating pain, respectively.

SECONDARY OUTCOMES:
The mean of back pain between two groups | Within 4 hours after TACE
  The patients were asked to describe their back pain and rate its severity by using the Numerical Rating Scale (NRS).To determine if there is any significant difference the two groups.
The mean of back pain in the experimental group | Within 4 hours after TACE
  To determine if there is any significant difference across the five-time periods in experimental group.
The mean of back pain in the control group | Within 4 hours after TACE
  To determine if there is any significant difference across the five-time periods in control group.
Vascular complication | Femoral puncture sites were assessed every hourly for the following 4 hours by researcher and a nurse.
  The hematoma in femoral access site or there is blood on the yarn roll were visually checked, its margin was marked by a marker and its size was measured by using measuring paper. (The area equal to a square that is 1 millimeter on each side).
Post embolization syndrome | Within 4 hours after TACE.
  This is a dichotomized variable. Various common symptoms were listed and checked off based on the patient's report.
Patients' satisfaction | Patient's satisfaction will be evaluated at the 4th hour.
  5-Point Likert Scale: with scores of 5, 4, 3, 2, and 1 indicating highly satisfied, satisfied, neutral, dissatisfied, and highly dissatisfied, respectively. Higher scores mean higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Tse-Pin Hsu, M.S.N., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chang KT, Liu CJ, Tsai HT, Hsu TP, Chen PT, Hu SH. Effects and safety of body positioning on back pain after transcatheter arterial chemoembolization in people with hepatocellular carcinoma: A randomized controlled study. Int J Nurs Stud. 2020 Sep;109:103641. doi: 10.1016/j.ijnurstu.2020.103641. Epub 2020 May 16. PMID 32535341